CLINICAL TRIAL: NCT00262041
Title: A Phase 2, Randomized, Single-blind, Controlled, Multicenter Study to Compare the Safety and Immune Response of One Dose of Novartis Meningococcal ACWY Conjugate Vaccine With the Safety and Immune Response of One Dose of Licensed Meningococcal ACWY Polysaccharide Vaccine Administered to Healthy Adolescents 11 to 17 Years of Age
Brief Title: Study of the Safety and Immune Response of a Meningococcal Conjugate Vaccine Administered to Healthy Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V59P6; BB-IND 11278
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Prevention of Meningococcal Disease

ARMS (3):
- MenACWY-CRM(Ad+) (Experimental): Subjects received one single dose of adjuvanted formulation of conjugate vaccine.
  Interventions: Biological: MenACWY-CRM conjugate vaccine, adjuvanted
- MenACWY-CRM(Ad-) (Experimental): Subjects received one single dose of unadjuvanted formulation of conjugate vaccine.
  Interventions: Biological: MenACWY-CRM conjugate vaccine, unadjuvanted
- MenACWY- PS (Active Comparator): Subjects received one single dose of the polysaccharide vaccine.
  Interventions: Biological: MenACWY polysaccharide vaccine

INTERVENTIONS:
Biological: MenACWY-CRM conjugate vaccine, adjuvanted
  Arms: MenACWY-CRM(Ad+)
Biological: MenACWY-CRM conjugate vaccine, unadjuvanted
  Arms: MenACWY-CRM(Ad-)
Biological: MenACWY polysaccharide vaccine
  Arms: MenACWY- PS

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of Novartis Meningococcal ACWY Conjugate Vaccine in comparison to licensed meningococcal polysaccharide vaccine administered to healthy adolescents ages 11 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents between and including 11-17 years of age, who provide written informed consent

Exclusion Criteria:

* Subjects with a previous or suspected disease caused by N. meningitidis; or previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s); Any serious acute, chronic or progressive disease

Ages: 11 Years to 17 Years | Sex: All
Age Groups: Child
Enrollment: 524 (Actual)
Dates: Start 2004-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Director — Novartis
Locations (3):
- United States (3):
  - Rochester, Minnesota
  - Pittsburgh, Pennsylvania
  - Seattle, Washington

REFERENCES:
- [Background] Jackson LA, Jacobson RM, Reisinger KS, Anemona A, Danzig LE, Dull PM. A randomized trial to determine the tolerability and immunogenicity of a quadrivalent meningococcal glycoconjugate vaccine in healthy adolescents. Pediatr Infect Dis J. 2009 Feb;28(2):86-91. doi: 10.1097/INF.0b013e31818a0237. PMID 19116603
- [Derived] Jacobson RM, Jackson LA, Reisinger K, Izu A, Odrljin T, Dull PM. Antibody persistence and response to a booster dose of a quadrivalent conjugate vaccine for meningococcal disease in adolescents. Pediatr Infect Dis J. 2013 Apr;32(4):e170-7. doi: 10.1097/INF.0b013e318279ac38. PMID 23114372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Seattle, Washington; Pittsburgh, Pennsylvania; Rochester, Minnesota.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenACWY-PS: Subjects received one single dose of the MenACWY polysaccharide vaccine.
Period: Overall Study
Arm/Group | MenACWY-CRM(Ad+) | MenACWY-CRM(Ad-) | MenACWY-PS
Started | 164 | 151 | 209
Completed | 162 | 147 | 203
Not Completed | 2 | 4 | 6
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 5
Not completed — Unable to classify | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MenACWY-PS - Stage 1: Subjects received a single of MenACWY polysaccharide vaccine on day 1 (Stage 1 - 1:1 randomization scheme).
- MenACWY-PS -Stage 2: Subjects received a single dose of MenACWY polysaccharide vaccine (Stage 2 - 4:1 MenACWY-CRM:MenACWY-PS randomization scheme).
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM(Ad+) | MenACWY-CRM(Ad-) | MenACWY-PS - Stage 1 | MenACWY-PS -Stage 2 | Total
Number analyzed (Participants) | 164 | 151 | 170 | 39 | 524
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.9) | 14.1 (1.8) | 14.2 (1.8) | 14.2 (2.0) | 14.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 62 | 70 | 11 | 209
  Male | 98 | 89 | 100 | 28 | 315

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With N.Meningitidis Human Serum Bactericidal Activity (hSBA) Titers≥ 1:4, After One Dose of Either MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, or MenACWY-PS Vaccine
Description: Immune response of a single dose of MenACWY-CRM conjugate vaccine, with adjuvant or without adjuvant compared to that of one dose of MenACWY polysaccharide (PS) vaccine, one month after administration to subjects aged 11 to 17 years, as measured by the percentage of subjects with hSBA titers >1:4 directed against N meningitidis serogroups A, C, W and Y
Time Frame: 1 month after vaccination
Population: Analysis was done on the per-protocol population i.e all subjects who received all the relevant doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol violation.
Measure: Number (95% Confidence Interval); unit: Percentages Of Subjects
Arm/Group | MenACWY-CRM(Ad+) | MenACWY-CRM(Ad-) | MenACWY-PS
Number analyzed (Participants) | 161 | 148 | 179
Percentages Of Subjects
  MenA (N=158,148,179) | 87 [80 to 92] | 84 [77 to 89] | 46 [38 to 53]
  MenC (N=161,148,177) | 93 [87 to 96] | 88 [81 to 93] | 71 [64 to 78]
  MenW (N=161,146,173) | 98 [94 to 99] | 95 [90 to 98] | 88 [83 to 93]
  MenY (N=159, 147,177) | 97 [93 to 99] | 96 [91 to 98] | 84 [77 to 89]
Statistical Analysis 1: Comparison: MenACWY-CRM(Ad+) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad+ vaccine group against serogroup A compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad+ vaccine against the serogroup A was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: MenACWY-CRM(Ad-) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad- vaccine group against serogroup A compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad- vaccine against the serogroup A was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: MenACWY-CRM(Ad+) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad+ vaccine group against serogroup C compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad+ vaccine against the serogroup C was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: MenACWY-CRM(Ad-) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad- vaccine group against serogroup C compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad- vaccine against the serogroup C was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p = 0.003, Chi-squared
Statistical Analysis 5: Comparison: MenACWY-CRM(Ad+) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad+ vaccine group against serogroup W compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad+ vaccine against the serogroup W was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p < 0.001, Chi-squared
Statistical Analysis 6: Comparison: MenACWY-CRM(Ad-) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad- vaccine group against serogroup W compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad- vaccine against the serogroup W was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p = 0.071, Chi-squared
Statistical Analysis 7: Comparison: MenACWY-CRM(Ad+) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad+ vaccine group against serogroup Y compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad+ vaccine against the serogroup Y was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p < 0.001, Chi-squared
Statistical Analysis 8: Comparison: MenACWY-CRM(Ad-) vs MenACWY-PS; To demonstrate non-inferiority of percentages of subjects with hSBA titer ≥ 1:4 who received MenACWY Ad- vaccine group against serogroup Y compared with that of MenACWY PS vaccine; Test type: Non-Inferiority or Equivalence — Non-inferiority of MenACWY Ad- vaccine against the serogroup Y was assessed to that of the MenACWY PS vaccine if the lower limit of the two-sided 95% CI around the difference in proportions was greater than -10%; p < 0.001, Chi-squared

2. Secondary Outcome: hSBA Geometric Mean Titers (GMT) After One Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant or MenACWY-PS Vaccine
Description: Immune response of one dose of MenACWY-CRM conjugate vaccine, with adjuvant or without adjuvant or MenACWY-PS vaccine, one month after administration in subjects 11 to 17 years of age, as measured by hSBA geometric mean titers (GMTs) against N meningitidis serogroups A, C, W, and Y.
Time Frame: 1 month after vaccination
Population: Analysis was done on per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM(Ad+) | MenACWY-CRM(Ad-) | MenACWY-PS
Number analyzed (Participants) | 161 | 148 | 179
Titers
  MenA (N=158, 148, 179) | 34 [26 to 43] | 34 [26 to 44] | 6.97 [5.51 to 8.82]
  MenC (N=161, 148, 177) | 69 [48 to 100] | 58 [39 to 85] | 30 [22 to 43]
  MenW (161, 146, 173) | 61 [49 to 75] | 49 [39 to 62] | 30 [24 to 37]
  MenY (159,147,177) | 112 [85 to 147] | 100 [75 to 133] | 34 [27 to 44]

3. Secondary Outcome: Percentages of Subjects With hSBA Titers≥ 1:4, After One Dose Of Either MenACWY-CRM(Ad-) or MenACWY-PS Vaccine
Description: Immune response of one dose of MenACWY-CRM(Ad-) compared to that of one dose of MenACWY polysaccharide(MenACWY-PS) vaccine, 12 months after administration to subjects aged 11 to 17 years, as measured by the percentage of subjects with human complement serum bactericidal activity (hSBA) titers≥1:4 against N meningitidis serogroups A, C, W, and Y. The endpoint point compares only data of unadjuvanted formulation of the conjugate vaccine to the polysaccharide vaccine.
Time Frame: 12 months after vaccination
Population: Analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentages Of Subjects
Arm/Group | MenACWY-CRM(Ad-) | MenACWY-PS
Number analyzed (Participants) | 140 | 149
Percentages Of Subjects
  MenA (N=140, 149) | 36 [28 to 44] | 44 [36 to 53]
  MenC (N=140, 147) | 86 [79 to 91] | 69 [61 to 76]
  MenW (N=138, 141) | 95 [90 to 98] | 72 [63 to 79]
  MenY (N=139, 147) | 87 [80 to 92] | 63 [54 to 70]

4. Secondary Outcome: hSBA Geometric Mean Titers (GMT) After One Dose Of Either MenACWY-CRM(Ad-) or MenACWY-PS Vaccine
Description: Immune response of one dose of MenACWY-CRM(Ad-) conjugate vaccine compared with that of MenACWY-PS vaccine, 12 months after administration in subjects 11 to 17 years of age, as measured by hSBA geometric mean titers (GMTs) against N meningitidis serogroups A, C, W, and Y.The endpoint compares only data of unadjuvanted formulation of the conjugate vaccine to the polysaccharide vaccine.
Time Frame: 12 months after vaccination
Population: Analysis was done on PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM(Ad-) | MenACWY-PS
Number analyzed (Participants) | 140 | 149
Titers
  MenA(N=140, 149) | 4.24 [3.35 to 5.38] | 5.65 [4.54 to 7.03]
  MenC (N=140, 147) | 28 [19 to 41] | 26 [18 to 37]
  MenW (N=138, 141) | 40 [31 to 52] | 17 [13 to 22]
  MenY (N=139, 147) | 30 [22 to 41] | 13 [9.49 to 17]

5. Secondary Outcome: Numbers of Subjects 11 to 17 Years of Age Who Reported Solicited Local and Systemic Adverse Events After the Vaccination
Description: Safety was assessed as the number of subjects 11 to 17 years of age who reported solicited local and systemic adverse events from day 1 up to and including day 7 after the vaccination of either MenACWY-CRM conjugate vaccine, with adjuvant or without adjuvant or MenACWY-PS vaccine.
Time Frame: Day 1 to Day 7
Population: Analysis was done on safety dataset - subjects who received at least one study dose and had Post baseline safety data.
Measure: Number; unit: Subjects
Groups:
- MenACWY-PS - Stage 1: Subjects received a single of MenACWY polysaccharide vaccine on day 1 (Stage 1)
- MenACWY-PS -Stage 2: Subjects received a single dose of MenACWY polysaccharide vaccine (Stage 2)
Arm/Group | MenACWY-CRM(Ad+) | MenACWY-PS - Stage 1 | MenACWY-CRM(Ad-) | MenACWY-PS -Stage 2
Number analyzed (Participants) | 164 | 170 | 151 | 39
Subjects
  Any Local | 103 | 102 | 107 | 24
  Injection Site Pain | 92 | 95 | 81 | 19
  Injection Site Erythema | 33 | 28 | 57 | 11
  Injection Site Induration | 22 | 15 | 34 | 8
  Any Systemic | 72 | 79 | 85 | 23
  Chills | 12 | 10 | 24 | 6
  Nausea | 15 | 20 | 22 | 0
  Malaise | 19 | 14 | 23 | 7
  Myalgia | 25 | 25 | 35 | 5
  Arthralgia | 13 | 5 | 12 | 2
  Headache | 60 | 63 | 62 | 19
  Fever ≥ 38°C | 2 | 3 | 1 | 1
  Any Other | 44 | 45 | 40 | 14
  Analgesic/Antipyretic Med Used | 44 | 45 | 39 | 14
  Stayed home Due to a reaction | 2 | 2 | 6 | 2

ADVERSE EVENTS:
Time Frame: All solicited adverse events (AEs) were collected upto day 7 after each vaccination.
Description: All AEs through day 7 and/or all serious adverse events (SAEs) and/or AEs requiring a physician visit and/or resulting in premature withdrawal from the study from day 1 to study termination (day 360).
Arm/Group | MenACWY-CRM(Ad+) | MenACWY-CRM(Ad-) | MenACWY-PS - Stage 1 | MenACWY-PS -Stage 2
Serious Adverse Events (participants affected / at risk) | 4/164 | 2/151 | 5/170 | 2/39
Other Adverse Events (participants affected / at risk) | 123/164 | 126/151 | 128/170 | 31/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM(Ad+) (N=164) | MenACWY-CRM(Ad-) (N=151) | MenACWY-PS - Stage 1 (N=170) | MenACWY-PS -Stage 2 (N=39)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis Pharyngeal (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arachnoid Cyst (Nervous system disorders) | 0 | 0 | 1 | 0
Hallucination, Auditory (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM(Ad+) (N=164) | MenACWY-CRM(Ad-) (N=151) | MenACWY-PS - Stage 1 (N=170) | MenACWY-PS -Stage 2 (N=39)
Nausea (Gastrointestinal disorders) | 15 | 22 | 20 | 0
Chills (General disorders) | 12 | 24 | 10 | 6
Injection Site Erythema (General disorders) | 33 | 57 | 28 | 11
Injection Site Induration (General disorders) | 22 | 34 | 15 | 8
Injection Site Pain (General disorders) | 92 | 81 | 95 | 19
Malaise (General disorders) | 20 | 23 | 14 | 7
Pharyngitis (Infections and infestations) | 6 | 2 | 4 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 12 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 12 | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 35 | 25 | 5
Headache (Nervous system disorders) | 60 | 62 | 63 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days